Title: A Study of Mobile Medical Supportive Care Program for Family Caregivers

With Dementia Combined With Diabetes

**Identifiers**: NCT06785857

Unique Protocol ID: K2021-05-024

Date: 2021-5-1

**Informed Consent** 

Dear uncle/aunt:

Greetings!

I am a graduate student of the School of Nursing, Fujian Medical University, and I am

" Development and application of nursing currently working on the project

intervention technology system for cognitive impairment in the elderly". The main

purpose of this study is to explore whether effective supportive care can effectively

improve the burden of care of dementia combined with diabetes mellitus caregivers.

You are invited to take part in this study, which will last 12 weeks. If you are willing

to participate, you will be assessed for caregiving burden.

SPECIAL NOTE: We guarantee that all information about your participation in the

study is confidential and that this investigation will not cause any harm to you or your

family. Therefore, the evaluation and examination are provided free of charge, and

you are free to choose to participate or decline this study, and also have the right to

withdraw from this study at any time.

If you are aware of the above information, please sign the Informed Consent section.

Again, thank you very much for your support and cooperation!

Researcher:

Informed on: (month and year)

| I have been | informed | of the | purpose | and | process | of this | study | and | have | the | right | to |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| withdraw freely, and I voluntarily participate in this study. | | | | | | | | | | | | |

Participant Signature:

Date: